CLINICAL TRIAL: NCT03562442
Title: Leibniz Association Senate Board of Competition (SAW) Lung Microbiome Study
Brief Title: SAW Lung Microbiome Study in Smokers and Never-smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center Borstel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SAW Lungenmikrobiom-Studie
Record Dates: First submitted 2018-05-26; First posted 2018-06-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation; Chronic Obstructive Pulmonary Disease (COPD); Healthy; Microbial Colonization
MeSH Terms: conditions — Smoking Cessation; Pulmonary Disease, Chronic Obstructive; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Two groups are recruited in parallel (A) Smokers who quit smoking (Visit 1 before cessation, Visit 2 six weeks after cessation) (B) Never-smokers (Visit 1 only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Experimental): Healthy caucasian smokers who are willing to quit smoking are investigated before cessation (Visit 1) and 6 weeks after cessation (Visit 2).
  Intervention: Smoking cessation
  Interventions: Behavioral: Smoking cessation
- Never-Smokers (No Intervention): Healthy caucasian volunteers who never smoked are investigated once only (Visit 1)

INTERVENTIONS:
Behavioral: Smoking cessation — Smoking cessation with or without professional / medical support
  Arms: Smokers

SUMMARY:
The trial aims to analyse changes in the microbiome of the lower airways after smoking cessation. Microbiome analyses (upper airway swabs, bronchoalveolar lavage, transbronchial brushing) are conducted in smokers before and 6 weeks after smoking cessation. Never smokers serve as a control group and undergo the same sampling procedures once.

DETAILED DESCRIPTION:
The trial aims to analyze changes in the microbiome of the lower airways after smoking cessation. Microbiome analyses (upper airway swabs, bronchoalveolar lavage, transbronchial brushing) are conducted in healthy (and willing to quit) smokers before and 6 weeks after smoking cessation. Never smokers serve as a control group and undergo the same sampling procedures once.

Demographic and clinical data of the study subjects are obtained, aiming for homogeneous groups. All personal data are encrypted according to the standard operating procedures of the study site. Pharyngeal and deep nasal swabs are taken.

To avoid contamination of the lower airways from the oropharynx through the bronchoscope, standardized procedures are established according to the German guidelines for bronchoscopy. Before bronchoscopy, the endoscope is flushed with sterile saline which is analyzed for 16S ribosomal RNA (rRNA) to control for residual contaminating bacterial desoxyribonucleic acid (DNA). A 300ml bronchoalveolar lavage with warm normal saline solution is taken from the middle lobe. Three covered and "microbiologically protected" bronchial brushings are obtained from the right upper lobe. This sterile brush is sealed in wax and pushed through the wax just before taking the brushing. All samples are immediately frozen and stored at -80°C until further analyses. For cultivations, samples are kept at 4°C and rapidly processed.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette consumption of at least five cigarettes per day
* Caucasian ethnicity

Exclusion Criteria:

* Continous passive smoking exposure
* Systemic steroid therapy during the previous month
* Chronic lung disease (exception COPD stage Global Initiative on Lung Disease (GOLD) 0/I/II)
* Diabetes mellitus
* Pregnancy or breast feeding
* active tuberculosis (currently or previously)
* respiratory infection in the previous month
* antibiotic therapy in the previous two months
* immunosuppression
* malignancy
* interstitial lung disease
* rheumatic disease with lung manifestation
* member of a collaborative group of the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in microbiome pattern in smokers after smoking cessation | 6 Weeks
  Number of bacteria genera in the lung identified by 16S rRNA and bacterial culture

SECONDARY OUTCOMES:
Smoking cessation rates | 6 weeks
  Percentage of sustained smoking cessation
Smoking cessation rates | 6 months
  Percentage of sustained smoking cessation
Lung microbiome in never-smokers | 0 days
  Number of bacteria genera in the lung identified by 16S rRNA and bacterial culture

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center Borstel, Borstel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfeiffer S, Herzmann C, Gaede KI, Kovacevic D, Krauss-Etschmann S, Schloter M. Different responses of the oral, nasal and lung microbiomes to cigarette smoke. Thorax. 2022 Feb;77(2):191-195. doi: 10.1136/thoraxjnl-2020-216153. Epub 2021 Aug 13. PMID 34389656